CLINICAL TRIAL: NCT05865158
Title: CardioSafe Plus: A Platform for Telerehabilitation and Monitoring of Patients With Heart Problems.
Brief Title: CardioSafe+: A Platform for Telerehabilitation and Monitoring of Patients With Heart Problems
Acronym: CardioSafe+
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Beatriz-María Bermejo-Gil, Assistant professor doctor, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CardioSafe+
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Institionalized group (Experimental): Group of institutionalized people with chronic cardiovascular diseases.
  Interventions: Other: Home-based exercises
- Community-dwelling group (Experimental): Group of community-dwelling people with chronic cardiovascular diseases.
  Interventions: Other: Home-based exercises

INTERVENTIONS:
Other: Home-based exercises — Home-based exercises proposed through the CardioSafe+ platform, guided by therapists specialized in cardiovascular disorders, who will try to adapt the sessions to each participant.

SUMMARY:
The use of telerehabilitation seems to be effective in managing complications after suffering a cardiovascular pathology. The use of the CardioSafe+ digital platform is suggested for the management of these complications. For this reason, an intervention will be carried out to determine the effectiveness of this platform. A total of 60 participants will be recruited to carry out a home-exercise intervention through CardioSafe+ for 6 weeks. Maximun respiratory pressures, exertion capacity, and subjective sensation of exertion will be assessed.

DETAILED DESCRIPTION:
This intervention seeks to determine the effectiveness of the CardioSafe+ digital platform in aiding individuals recovering from cardiovascular pathologies. By involving a group of 60 participants in a structured six-week home-exercise program using the CardioSafe+ platform, the objective is to measure and evaluate various factors related to their physical well-being and recovery.

Key components to be evaluated include:

Maximal Respiratory Pressures: This involves measuring the maximum force generated during inspiration and expiration, which can indicate respiratory muscle strength and function.

Exertion Capacity: The assessment aims to gauge the participants' ability to engage in physical activities, potentially reflecting improvements in overall cardiovascular fitness and endurance.

Subjective Sensation of Exertion: This component involves understanding how the participants perceive and rate their own exertion during exercises, contributing to insights about their subjective experience and effort perception.

The intervention's objective is to collect data on these parameters before and after the six-week exercise program utilizing the CardioSafe+ digital platform. This data will help determine the effectiveness of the platform in aiding individuals recovering from cardiovascular pathologies and could provide valuable insights for further implementing tele-rehabilitation in managing such health complications.

ELIGIBILITY:
Inclusion Criteria:

* People who present a cardiovascular pathology with more than one year of evolution.
* To be in a stable medical situation.
* To have access to technological resources and knowledge for their use.

Exclusion Criteria:

* People who present any contraindication established for carrying out physical activity.
* People who present insufficient capacity to understand and obey the instructions offered by the researchers, both in the evaluation and in the intervention.
* People who have a cardiac pathology with obvious fluctuations in the course of the disease.
* The presence of an acute episode of the disease during the intervention period.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-20 (Actual); Primary Completion 2024-06-22 (Estimated); Study Completion 2024-06-22 (Estimated)

PRIMARY OUTCOMES:
Maximum inspiratory pressure by spirometry | 6 weeks
  Value of the maximum inspiratory capacity in mm of H2O.
Maximum expiratory pressure by spirometry | 6 weeks
  Value of the maximum expiratory capacity in mm of H2O.
Borg Rating of Perceived Exertion Scale | 6 weeks
  Scale of perceived subjective effort in which it is valued with a score of 0 to 10, subjectively. Started from 0 where your breathing is causing you no difficulty at all and progresses through to number 10 where your breathing difficulty is maximal.
2 minute stationary walk test | 6 weeks
  Effort test in which the participant is asked to lift their knees for 2 minutes and the number of times is counted. Based on that number, the percentile in which the person is based on their age and sex is calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz María Bermejo Gil, Principal Investigator — University of Salamanca
Locations (1):
- Beatriz María Bermejo Gil, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No
Los datos de los participantes se trataran segun la Ley Orgánica 3/2018, de 5 de diciembre, de Protección de Datos Personales y garantía de los derechos digitales.